CLINICAL TRIAL: NCT01306539
Title: Neuropsychiatric Effects of Deep Brain Stimulation in Patients With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Adam Aron, Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: HSC-07-4849
Record Dates: First submitted 2011-02-28; First posted 2011-03-02 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Parkinson's Disease
Keywords: deep brain stimulation; subthalamic nucleus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deep Brain Stimulation (Experimental): Parkinson's patients with deep brain stimulation in the subthalamic nucleus.
  Interventions: Procedure: Stimulation of the subthalamic nucleus

INTERVENTIONS:
Procedure: Stimulation of the subthalamic nucleus — Stimulation is delivered to the subthalamic nucleus at experimentally prescribed settings.

SUMMARY:
Stimulation of the subthalamic nucleus will have effects on various aspects of neuropsychiatric function.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with idiopathic Parkinson's disease that meet criteria for treatment of their disease with STN-DBS. Participants will be selected for this study without regard for age (provided they are older than 18), gender or ethnic background.
* Participants must have undergone subthalamic nucleus DBS surgery and be receiving treatment at the Scripps Clinic in La Jolla, CA

Exclusion Criteria:

* Patients under 18 years old.
* Patients with mini-mental status scores below 26/30.
* Patients with known psychiatric disease.
* Patients who are too infirm, demented or dysarthric to clearly understand the consenting process, task instructions, or to communicate verbally regarding participation or non-participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
behavioral task performance | 1 to 2 hours
  Participants will complete behavioral tasks at each of three visits to assess the effects of stimulation settings on task performance. At each research visit, behavior will be assessed beginning at 1 hour after the stimulation is adjusted to the experimental settings. Stimulation settings will be returned to each patient's treatment levels at the culmination of each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Aron, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- Scripps Clinic Torrey Pines, La Jolla, California, United States

REFERENCES:
- [Result] Greenhouse I, Gould S, Houser M, Hicks G, Gross J, Aron AR. Stimulation at dorsal and ventral electrode contacts targeted at the subthalamic nucleus has different effects on motor and emotion functions in Parkinson's disease. Neuropsychologia. 2011 Feb;49(3):528-34. doi: 10.1016/j.neuropsychologia.2010.12.030. Epub 2010 Dec 22. PMID 21184765